CLINICAL TRIAL: NCT05363124
Title: Evaluation of Mobile App to Assist in Pediatric Triage in a Pediatric Emergency Department
Brief Title: Evaluation of Mobile App to Assist in Pediatric Triage
Acronym: PEWSAPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-HPNCL-05
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Pediatric Triage in a Pediatric Emergency Department

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEWS calculation (Experimental): PEWS calculation by parents using AI-based smartphone app PEWS calculation by nurse using conventional procedure
  Interventions: Other: PEWS calculation by parents using AI-based smartphone app; Other: PEWS calculation by nurse using conventional procedure

INTERVENTIONS:
Other: PEWS calculation by parents using AI-based smartphone app — After patient registration, the patient will be installed in the nursing office with one of his parents . After screening a potential life-threatening patient for which treatment would be started first of all, the nurse will collect the signed parental consent for participating to the study. Explanations will be given to the parents regarding the use of the application and the way to calculate the PEWS through a very brief and standardized education. Parents should then proceed to the calculation of PEWS, as far as possible before the intervention of the nurse, using the Caducy® appl with a smartphone dedicated to the study .
Other: PEWS calculation by nurse using conventional procedure — After patient registration, the patient will be installed in the nursing office with one of his parents . After screening a potential life-threatening patient for which treatment would be started first of all, the nurse will collect the signed parental consent for participating to the study. the nurse proceed to the calculation of PEWS in blind of parents and to triage process by priorityzing patient in 5 level of gravity (from 1-vital emergency to 5-nonurgent patient). If the medical examination was not proceeded directly after the triage process, nurses were asked to proceed a new triage if the optimal delay of the medical examination was passed.

SUMMARY:
Each ED manages a wide variety of pathologies ranging from a simple general consultation to a life-threatening emergency. Patients require prioritization and triaging as soon as they reach the ED and cannot be seen purely in the order of arrival. This triage is mostly carried out by a nurse at the triage zone who must quickly identify high-emergency patients requiring immediate care and organize their care pathway. The triage nurse uses a decision support tool known as a triage tool.

In 2000, the PED of the University Hospital of Nice (France) created a 5-level pediatric triage tool - the pediaTRI - based on clinical items of inspection, interview, and analysis of vital signs.

In a pediatric ED (PED) setting, a high-level emergency corresponds to a child presenting an immediate life-threatening risk that could lead to cardio-respiratory arrest or a related emergency, and thus requires rapid intervention. These patients, for whom a Level 1 or 2 is usually assigned by commonly used pediatric triage tools, can also be screened using warning scores that are predictive of clinical deterioration within 24 hours after visiting the PED. Among them, the Pediatric Early Warning System (PEWS) system, created in 2001, is considered to be efficient, easy to use, and reliable. According to the literature, the optimal cutoff level to calculate the sensitivity and specificity for admission to an ICU, defined as a high-level emergency, is ≥ 4/9. Vitals signs used to calculate the PEWS are usually collected by the nurse at the triage zone. However, new technology such as mobile application may be also used to capture those vital signs (i-Virtual).

Since the parameters of the PEWS system may be evaluate by parents using the application, the investigators want to analyze their ability to assess the level of severity of their children by scoring PEWS in a pediatric emergency department using the mobile application Caducy® (i-Virtual)

DETAILED DESCRIPTION:
The number of visits to emergency departments (ED) has been rising steadily for both adult and pediatric patients over the past decades. resulting in an increase in waiting and care times. Each ED manages a wide variety of pathologies ranging from a simple general consultation to a life-threatening emergency. However, overcrowding in the ED as well as difficulties in monitoring patients waiting for clinical examination, can endanger patient safety. Patients require prioritization and triaging as soon as they reach the ED and cannot be seen purely in the order of arrival. An ideal triage system should be able to identify those who require immediate care (high-level emergency) from those who can wait or those who will not require emergency care (intermediate- to low-level emergency). This triage is mostly carried out by a nurse at the triage zone who must quickly identify high-emergency patients requiring immediate care and organize their care pathway. The triage nurse uses a decision support tool known as a triage tool.

In France, there is no gold standard in pediatric triage and each hospital uses their own "home-made" triage system. In 2000, the PED of the University Hospital of Nice (France) created a 5-level pediatric triage tool - the pediaTRI - based on clinical items of inspection, interview, and analysis of vital signs. In a pediatric ED (PED) setting, a high-level emergency corresponds to a child presenting an immediate life-threatening risk that could lead to cardio-respiratory arrest or a related emergency, and thus requires rapid intervention. These patients, for whom a Level 1 or 2 is usually assigned by commonly used pediatric triage tools, can also be screened using warning scores that are predictive of clinical deterioration within 24 hours after visiting the PED. Among them, the Pediatric Early Warning System (PEWS) system, created in 2001, is considered to be efficient, easy to use, and reliable. The PEWS system is based on three main components each given a 3-point rating as follows: (a) behavior and early signs of shock, recognizable and assessable by the parents; (b) skin tone and capillary refill time to assess the cardiovascular system; (c) and respiratory rate and oxygen dependence to assess the respiratory system. According to the literature, the optimal cutoff level to calculate the sensitivity and specificity for admission to an ICU, defined as a high-level emergency, is ≥ 4/9. Vitals signs used to calculate the PEWS are usually collected by the nurse at the triage zone. However, new technology such as mobile application may be also used to capture those vital signs (i-Virtual).

Since the parameters of the PEWS system may be evaluate by parents using the application, the investigators want to analyze their ability to assess the level of severity of their children by scoring PEWS in our pediatric emergency department using the mobile application Caducy® (i-Virtual).

ELIGIBILITY:
Inclusion Criteria:

* patients under 18
* visited the PED of Lenval Children's Hospital for medical reason
* Parental consent signed

Exclusion Criteria:

* Patients visited the PED of Lenval Children's Hospital for a reason other than medical
* A sign (s) of vital distress
* Patients who were called back,
* Patients treated in prehospital care,
* Patients who left without an assigned triage level
* Non-French speaking parents

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pediatric Early Warning System (PEWS) calculated by parent using smartphone app | at inclusion
  The Pediatric Early Warning System (PEWS) is based on three main components each given a 3-point rating as follows: (a) behavior and early signs of shock, recognizable and assessable by the parents; (b) skin tone and capillary refill time to assess the cardiovascular system; (c) and respiratory rate and oxygen dependence to assess the respiratory system.
  the PEWS score is calculated by parent using smartphone app and
  According to the score, patients will be classified as follows:
  * PEWS [0-2] = no risk
  * PEWS[3-4] = moderate risk
  * PEWS [5-9] = High risk
Pediatric Early Warning System calculated by nurse | at inclusion
  the PEWS score is calculated by nurse using conventional procedure. he Pediatric Early Warning System (PEWS) is based on three main components each given a 3-point rating as follows: (a) behavior and early signs of shock, recognizable and assessable by the parents; (b) skin tone and capillary refill time to assess the cardiovascular system; (c) and respiratory rate and oxygen dependence to assess the respiratory system.
  According to the score, patients will be classified as follows:
  * PEWS [0-2] = no risk
  * PEWS[3-4] = moderate risk
  * PEWS [5-9] = High risk

SECONDARY OUTCOMES:
PEWS calculated by parents after triage process | until 240 minutes maximum from inclusion
  PEWS is calculated again by parent using smartphone app If the medical examination was not proceeded directly after the triage process, nurses were asked to proceed a new triage of the patient if the optimal delay of the medical examination was passed. The delays after which a new triage process should be performed by the nurse are defined according to the triage level given by the nurse using the triage tool as follows:
  * Level 1: < 5 min
  * Level 2: < 20 min
  * Level 3: <60 min
  * Level 4: <120 min
  * Level 5: < 240 min
PEWS calculated by nurse after triage process | until 240 minutes maximum from inclusion
  PEWS is calculated again by nurse If the medical examination was not proceeded directly after the triage process
PEWS calculated by doctor | until 4 hours from inclusion
  PEWS is calculated by the doctor before the medical examination.
Agreement between PEWS and final orientation | through study completion, an average of 6 months
  Agreement (yes/no) between parents using Artificial Intelligent (AI)-based smartphone app and the nurse will be evaluated at the first and the last assessment of PEWS according to the final orientation as follows: discharged, hospitalization, operating room, intensive care unit
Agreement between PEWS and group of chief complaint at the triage | through study completion, an average of 6 months
  Agreement (yes/no) between parents using AI-based smartphone app and the nurse will be evaluated at the first assessment of PEWS according to the group of chief complaint at the triage as follows: medical complaints (categorized as: ear, nose and throat (ENT), pulmonary, cardiovascular, neurology, digestive, urology-nephrology, gynecology, dermatology, endocrinology-metabolism, infectious diseases, rheumatology and pain, hematology, poisoning, and others), surgical complaints (categorized as head and neck trauma, upper and lower limb trauma, trauma of the trunk-pelvis-urogenital apparatus, burns, and others).
Agreement between PEWS and diagnosis | through study completion, an average of 6 months
  Agreement between parents using AI-based smartphone app and the nurse will be evaluated at the first assessment of PEWS according to the group of diagnosis as follows: medical diagnosis and surgical
Agreement between PEWS and day period | through study completion, an average of 6 months
  Agreement (yes/no) between parents using AI-based smartphone app and the nurse will be evaluated at the first assessment of PEWS according to the time when patients have been firstly triaged by the nurse, as follows: opened days and hours (from monday to Friday 08 am to 20pm and Saturday morning 08am to 12pm), on-call (out of the range of time and day defined previously)
Agreement between PEWS and patient age | through study completion, an average of 6 months
  Agreement (yes/no) between parents using AI-based smartphone app and the nurse will be evaluated at the first assessment of PEWS according to the age groups classified as follows: 0 - 27 days, 28 days - 3 months, 3 months - 1 year, 1 - 3 years, 3 - 7 years, 7 - 12 years, and 12 - 18 years
parental satisfaction | at the end of patient participation, an average of 3 hours
  assessment of parental satisfaction by Likert scale from 1 (totally useless) to 5 (totally useful)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France